CLINICAL TRIAL: NCT07291063
Title: A Phase I/II Study of Anti-PD-1/PD-L1 Antibodies in Combination With Gemcitabine and Cisplatin for Patients With Advanced Cholangiocarcinoma
Brief Title: Anti-PD-1/PD-L1 Antibodies Plus Gemcitabine and Cisplatin for Advanced CCA
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Y2024-752
Record Dates: First submitted 2025-12-02; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma; Gemcitabine; Cisplatin; Anti-PD-1/PD-L1 antibody
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Gemcitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chemotherapy plus Immunotherapy Combination
  Interventions: Drug: Anti-PD-1/PD-L1 antibody; Drug: Gemcitabine and Cisplatin Chemotherapy

INTERVENTIONS:
Drug: Anti-PD-1/PD-L1 antibody — Anti-PD-1/PD-L1 Intravenous injection for at least 6 months
Drug: Gemcitabine and Cisplatin Chemotherapy — Gemcitabine and cisplatin Intravenous injection for at least 6 months

SUMMARY:
This study is a prospective, observational study designed to analyze the safety, tolerability, and efficacy of first-line treatment using the combination of gemcitabine and cisplatin plus anti-PD-1/PD-L1 antibodies for patients with advanced cholangiocarcinoma.

DETAILED DESCRIPTION:
This is a prospective cohort study of combination anti-PD-1/PD-L1 antibodies plus Gemcitabine and Cisplatin chemotherapy for adult patients (≥18) with advanced cholangiocarcinoma

Gemcitabine and Cisplatin (GC): This chemotherapy doublet has been the historical standard of care for advanced cholangiocarcinoma. It works by interfering with DNA synthesis and causing DNA cross-linking, leading to tumor cell apoptosis.

Anti-PD-1/PD-L1 antibodies: Immunotherapy (including pembrolizumab, durvalumab, envafolimab, tislelizumab, etc.) is designed to block the PD-1/PD-L1 immune checkpoint pathway, thereby reinvigorating T-cells to recognize and attack tumor cells. Recent pivotal trials (e.g., TOPAZ-1, KEYNOTE-966) have demonstrated that adding immunotherapy to GC chemotherapy significantly improves overall survival compared to chemotherapy alone.

This study aims to evaluate the real-world safety, tolerability, and clinical efficacy of this combination regimen in specific clinical practice settings for unresectable late-stage cholangiocarcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. ≥18 years old, male or female 2. Histologically or cytologically confirmed locally advanced or metastatic biliary tract cancer (including ICC, ECC, or GBC) that is not amenable to curative surgery or local therapies.

  3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 4. Patient has given written informed consent. 5. The function of important organs meets the requirements 6. Expected survival ≥12 weeks 7. Non-surgical sterilization or women of childbearing age need to use a medically-accepted contraceptive (such as an intrauterine device, contraceptive or condom) during the study period and within 3 months after the end of the study treatment period.

Exclusion Criteria:

* 1. The patient has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, thyroid Hyperfunction; patients with vitiligo; complete remission of asthma in childhood, can be included without any intervention after adulthood; asthma patients who require bronchodilators for medical intervention cannot be included); 2. The patient is using immunosuppressive agents or systemic hormonal therapy to achieve immunosuppressive purposes (agents amount > 10 mg / day of prednisone or other therapeutic hormones), and continue to use within 2 weeks before enrollment; 3. Have clinical symptoms or disease that are not well controlled; 4. Significant clinically significant bleeding symptoms or a clear bleeding tendency within 3 months prior to randomization; 5. Arterial/venous thrombosis in the first 6 months of randomization 6. According to the investigator, the patient has other factors that may affect the results of the study or lead to the termination of the study, such as alcohol abuse, drug abuse, other serious diseases (including mental illness) requiring combined treatment, and serious laboratory abnormalities.#with family or social factors, it will affect the safety of patients. 7. Known hypersensitivity to Gemcitabine, Cisplatin, or platinum-containing compounds; significant hearing impairment (grade ≥2) or peripheral neuropathy (grade ≥2) that contraindicates Cisplatin;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic biliary tract cancer diagnosed histologically or cytologically.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after last treatment dose
  Safety will be monitored by addressing and recording all adverse events (AEs), serious adverse events (SAEs) and specific laboratory abnormalities (worst grade). Toxicities will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0.
Objective response rate(ORR) | 5 years
  Evaluated by researchers based on the RECIST 1.1 standard
Progression free survival(PFS) | 5 years
  Evaluated by researchers based on the RECIST 1.1 standard
To the relief time (TOR) | Time Frame: 5 years
  Evaluated by researchers based on the RECIST 1.1 standard
Duration of relief(DOR) | 5 years
  Evaluated by researchers based on the RECIST 1.1 standard
Disease Control Rate (DCR) | Time Frame: 5 years
  Evaluated by researchers based on the RECIST 1.1 standard

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Result] Oh DY, Ruth He A, Qin S, Chen LT, Okusaka T, Vogel A, Kim JW, Suksombooncharoen T, Ah Lee M, Kitano M, Burris H, Bouattour M, Tanasanvimon S, McNamara MG, Zaucha R, Avallone A, Tan B, Cundom J, Lee CK, Takahashi H, Ikeda M, Chen JS, Wang J, Makowsky M, Rokutanda N, He P, Kurland JF, Cohen G, Valle JW. Durvalumab plus Gemcitabine and Cisplatin in Advanced Biliary Tract Cancer. NEJM Evid. 2022 Aug;1(8):EVIDoa2200015. doi: 10.1056/EVIDoa2200015. Epub 2022 Jun 1. PMID 38319896
- [Result] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Result] Kelley RK, Ueno M, Yoo C, Finn RS, Furuse J, Ren Z, Yau T, Klumpen HJ, Chan SL, Ozaka M, Verslype C, Bouattour M, Park JO, Barajas O, Pelzer U, Valle JW, Yu L, Malhotra U, Siegel AB, Edeline J, Vogel A; KEYNOTE-966 Investigators. Pembrolizumab in combination with gemcitabine and cisplatin compared with gemcitabine and cisplatin alone for patients with advanced biliary tract cancer (KEYNOTE-966): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2023 Jun 3;401(10391):1853-1865. doi: 10.1016/S0140-6736(23)00727-4. Epub 2023 Apr 16. PMID 37075781